CLINICAL TRIAL: NCT03461133
Title: Detection of Deteriorating Patients on Peripheral Surgical Wards by an Automated Notification System
Brief Title: Automated Early Warning Scoring on Surgical Normal Wards
Status: Completed | Type: Observational
Sponsor: University Hospital Carl Gustav Carus (Other)
Responsible Party: Principal Investigator, Axel R. Heller, Head of Emergency Services, University Hospital Carl Gustav Carus
Other Study IDs: DrePaSiNet
Record Dates: First submitted 2018-02-25; First posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Safety Issues; Emergencies
MeSH Terms: conditions — Emergencies | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Reference: All patients admitted to the participating surgical wards from 2015-01-01 to 2015-12-31
- Intervention: All patients admitted to the participating surgical wards from 2016-07-01 to 2017-06-30
  Interventions: Other: Intervention

INTERVENTIONS:
Other: Intervention — The emergency notification system is linked to a paging system to the surgeon in charge and to the Hospital Medical Emergency Team. Depending on individual Multiparameter Early Warning Score communication protocols are activated.
  Other Names: Automated early warning score and notification system
  Groups: Intervention

SUMMARY:
Establishment of early warning systems in hospitals was strongly recommended in recent guidelines to detect deteriorating patients early and direct them to adequate care. Upon meeting of predefined trigger criteria Medical Emergency Teams (MET) should be directed to these patients. The present study analyses the effect of introduction of an automated early warning and trigger system on two peripheral wards hosting a highly complex surgical patient cohort.

DETAILED DESCRIPTION:
The deployment of an electronic monitoring and notification system is accompanied by data acquisition over 12 months (intervention) using four routine databases: Hospital patient data management, anesthesia database, local data of the German Resuscitation Registry, and measurement logs of the automated patient monitoring and alert system (intervention period only). A preceding time period of 12 months served as control.

ELIGIBILITY:
Inclusion Criteria:

* Admission to one of the participating wards

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: General surgery, vascular surgery, thoracic surgery,
Sampling Method: Non-Probability Sample
Enrollment: 3827 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
In hospital cardiac arrests | on average 14 days per patient, cumulative over 12 months in each observed cohort
  Patient cardiac arrests during stay

CONTACTS AND LOCATIONS:
Overall Officials: Axel R. Heller, MD, Principal Investigator — University Hospital Dresden, GERMANY
Locations (1):
- University Hospital Dresden, Dresden, Germany

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared

REFERENCES:
- [Background] Pearse RM, Moreno RP, Bauer P, Pelosi P, Metnitz P, Spies C, Vallet B, Vincent JL, Hoeft A, Rhodes A; European Surgical Outcomes Study (EuSOS) group for the Trials groups of the European Society of Intensive Care Medicine and the European Society of Anaesthesiology. Mortality after surgery in Europe: a 7 day cohort study. Lancet. 2012 Sep 22;380(9847):1059-65. doi: 10.1016/S0140-6736(12)61148-9. PMID 22998715
- [Background] Ludikhuize J, Brunsveld-Reinders AH, Dijkgraaf MG, Smorenburg SM, de Rooij SE, Adams R, de Maaijer PF, Fikkers BG, Tangkau P, de Jonge E; Cost and Outcomes of Medical Emergency Teams Study Group. Outcomes Associated With the Nationwide Introduction of Rapid Response Systems in The Netherlands. Crit Care Med. 2015 Dec;43(12):2544-51. doi: 10.1097/CCM.0000000000001272. PMID 26317569
- [Background] Muller MP, Richter T, Papkalla N, Poenicke C, Herkner C, Osmers A, Brenner S, Koch T, Schwanebeck U, Heller AR. Effects of a mandatory basic life support training programme on the no-flow fraction during in-hospital cardiac resuscitation: an observational study. Resuscitation. 2014 Jul;85(7):874-8. doi: 10.1016/j.resuscitation.2014.03.046. Epub 2014 Mar 28. PMID 24686020
- [Background] Subbe CP, Duller B, Bellomo R. Effect of an automated notification system for deteriorating ward patients on clinical outcomes. Crit Care. 2017 Mar 14;21(1):52. doi: 10.1186/s13054-017-1635-z. PMID 28288655

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT03461133/Prot_SAP_000.pdf